CLINICAL TRIAL: NCT03897491
Title: Evaluation of the Feasibility of PD L 506 for Stereotactic Interstitial Photodynamic Therapy (iPDT) in Adult Patients With Newly Diagnosed Supratentorial IDH Wild-type Glioblastoma
Brief Title: PD L 506 for Stereotactic Interstitial Photodynamic Therapy of Newly Diagnosed Supratentorial IDH Wild-type Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: photonamic GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GL 01
Record Dates: First submitted 2019-03-19; First posted 2019-04-01 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interstitial photodynamic therapy (Experimental): 20 mg 5-aminolevulinic acid per kg body weight orally four hours (range 3,5-4,5 hours) before the induction of general anaesthesia.
  Interventions: Drug: 5-aminolevulinic acid

INTERVENTIONS:
Drug: 5-aminolevulinic acid — 5-aminolevulinic acid powder for oral solution

SUMMARY:
The trial is an open, multicenter, explorative, pilot phase II study in a small number of patients to assess safety and efficacy of stereotactic interstitial photodynamic therapy (iPDT) with PD L 506 in newly diagnosed supratentorial IDH wild-type glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven, newly diagnosed, supratentorial, unifocal, lobar located IDH wild-type glioblastoma according to the criteria of the 2016 WHO classification.
* Not safely and/or not completely resectable, lobar located, unifocal, supratentorial IDH wild-type glioblastomas with a largest diameter ≤ 40 mm (largest diameter of the contrast enhanced tumor, as defined by enhanced T1 MRI sequences) are eligible in case of corresponding tumor board re-estimations.
* Potentially completely resectable, lobar located, unifocal, supratentorial, IDH wild-type glioblastoma with a largest diameter ≤ 40 mm are eligible in case of both patient's informed preference in favour of iPDT and corresponding tumor board recommendations.
* Age 18 - 70 years
* Karnofsky Performance status (KPS) of ≥ 70 %
* Minimal life expectancy of 3 months.
* Patients eligible for radiotherapy plus concomitant and adjuvant chemotherapy with temozolomide: Adequate haematological function (Absolute neutrophil count (ANC) > 1.5 x 109/L, Platelet count > 100 x 109/L, Haemoglobin > 10 g/dL (may be transfused to maintain or exceed this level)).
* International normalized ratio (INR) or PT (secs) and activated partial thromboplastin time (aPTT) ≤ 1,5 times of the upper limit of normal in the laboratory where it was measured.
* Negative pregnancy test in fertile women
* For female and male patients of reproductive potential: Willingness to apply highly effective contraception (Pearl index <1) during the entire study.

Such methods include :

* combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

  * oral
  * intravaginal
  * transdermal
* progestogen-only hormonal contraception associated with inhibition of ovulation :

  * oral
  * injectable
  * implantable
* intrauterine device (IUD)
* intrauterine hormone-releasing system (IUS)
* bilateral tubal occlusion
* vasectomised partner
* sexual abstinence • Written informed consent has been signed and dated prior to or at the beginning of Visit -1

Exclusion criteria:

* Glioblastomas involving the basal ganglia, the corpus callosum, the primary motor cortex, the ventricular system, multifocal tumors, and those involving the brain stem and/or the cerebellum.
* Glioblastomas exceeding the 40 mm threshold in their largest diameter
* Simultaneous use of other potentially phototoxic substances (e.g. tetracyclines, sulfonamides, fluoroquinolones, hypericin extracts)
* Hypersensitivity against porphyrins
* Known diagnosis of porphyria
* Acute or chronic hepatic diseases (levels of ASAT, ALAT and/or gamma-GT more than 2.5 times the upper limit of normal in the laboratory where it was measured)
* Manifest renal diseases with renal dysfunction (serum creatinine level > 1.5 times of the upper limit of normal in the laboratory where it was measured)
* Severe, active co-morbidity:
* Unstable angina and/or congestive heart failure within the last 6 months
* Transmural myocardial infarction within the last 6 months
* History of stroke, cerebral vascular accident, or transient ischemic attack within 6 months
* Serious and inadequately controlled cardiac arrhythmia
* Significant vascular disease (e.g. aortic aneurysm)
* Evidence of bleeding diathesis or coagulopathy
* Acute bacterial or fungal infections
* Acute exacerbation of chronic obstructive pulmonary disease
* Hepatic insufficiency resulting in clinical jaundice and/or coagulopathy
* Acquired immune deficiency syndrome; note, however, that HIV testing is not required for study entry.
* Inability to undergo MRI (e.g., presence of a pacemaker)
* Known intolerance to study medication
* Dementia or psychic condition that might interfere with the ability to understand the study and thus give a written informed consent
* Simultaneous participation in another clinical study or participation in another clinical study in the 30 days directly preceding treatment or within 5 plasma half-life of the preceding study drug, whatever is longer.
* Pregnancy or breastfeeding
* In case of both complete absence of intra-operative fluorescence between any of the inserted light diffusers and absence of significant surgery-associated bleedings (i.e. light transmission is detectable between at least two of the inserted light diffusers), the tumor will be classified as 'fluorescence-negative tumor'. iPDT will however be performed. Regarding efficacy evaluation, patients with fluorescence-negative tumors will be excluded from PP-, but included in the ITT-evaluation, and will be evaluated regarding safety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of treatment-emergent Adverse Events (safety and tolerability) of iPDT with PD L 506 in adult patients with newly diagnosed supratentorial IDH wild-type glioblastoma. | 2 weeks
  The incidence of treatment-emergent Adverse Events (TEAEs) of CTC grades 3, 4 and 5 within two weeks following iPDT

SECONDARY OUTCOMES:
Progression-free survival rate at 12 months | 12 months
  Percentage of patients without tumor progression 12 months after iPDT
Overall survival rate at 12 months | 12 months
  Percentage of patients who are alive 12 months after iPDT
Progression-free survival | From date of iPDT until the date of first documented progression, up to 66 months
  Time until first tumor progression
Overall survival | From date of iPDT until the date of death from any cause, up to 66 months
  Time until death from any cause
MGMT promoter methylation status of the patient | Baseline
  Analytical results for MGMT promoter methylation status (methylated/unmethylated) in the respective tumor samples of each patient
Immune status of the patient | Baseline, 2 days, 2 weeks after iPDT and then every 3 months, up to 66 months
  Analytical results for immune parameters (PBMC, CD4+, CD8+) in the respective blood samples of each patient
Results of investigator's assessment of patient's physical condition using Karnofsky performance status scale | Baseline, 2 weeks after iPDT and then every 3 months, up to 66 months
  To determine patient's physical condition using Karnofsky performance status scale ranging from 0% (worst outcome) to 100% (best outcome)
Results of investigator's assessment of patient's mental condition using Mini-mental State Examination | Baseline, 2 weeks after iPDT and then every 3 months, up to 66 months
  To determine patient's mental condition using Mini-mental State Examination scale ranging from 0 (worst outcome) to 30 (best outcome)
Results of investigator's assessment of patient's mental condition using National Institutes of Health Stroke Scale | Baseline, 2 weeks after iPDT and then every 3 months, up to 66 months
  To determine patient's mental condition using National Institutes of Health Stroke Scale ranging from 0 (best outcome) to 34 (worst outcome)
Results of investigator's assessment of patient's condition using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life of Cancer Patients Questionnaire (QLQ-C30) together with the Brain module (BN20) | Baseline, 2 weeks after iPDT and then every 3 months, up to 66 months
  To determine patient's quality of life
Interstitial light transmittance and fluorescence data recorded | during iPDT treatment (up to 1 hour)
  To determine whether correlations exist between length of OS/PFS and spectral online-monitoring measurement results (transmission and fluorescence measurements)
Interstitial fluorescence data recorded | during iPDT treatment (up to 1 hour)
  To determine the rate of patients with fluorescence-negative tumors
Percentage of cylindrical diffusor laser probes without kinks, cracks etc. before and after iPDT for patients treated under protocol versions prior to V7.0 | Day 0 (Treatment day), directly before and after iPDT
  Assessing the safety and performance of the insertion of Cylindrical Diffusor Laser Probes into the brain for iPDT of brain tumors for patients treated under protocol versions prior to V7.0.
Percentage of guiding catheters without kinks, cracks etc. before and after iPDT | Day 0 (Treatment day), directly before and after iPDT
  Assessing the safety and performance of the insertion of guiding catheters into the brain for iPDT of brain tumors
Percentage of iPDT treatments in which the laser system works properly as planned. | Day 0 (Treatment day), directly after iPDT
  Assessing safety and performance of the laser system for iPDT of brain tumors.
Percentage of fibers/laser ports which show a maximum deviation in the output power of less than +/-10% to the pre-defined output power of 200 mW/cm diffusor length. | Day 0 (Treatment day), directly after iPDT
  Assessing safety and performance of the combination of ML7710i laser system and Cylindrical Diffusor Laser Probes for the iPDT of brain tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stummer, Prof. Dr., Principal Investigator — Universitätsklinikum Münster
Locations (3):
- Germany (3):
  - Uniklinik Köln, Cologne
  - Klinikum der Universität München, München
  - Universitätsklinikum Münster, Münster

IPD SHARING:
Plan to Share IPD: No